Participant Informed Consent for Clinical Research

# Study title for participants: Examinations of Tissue from Ablated Malignant Liver Metastases as Predictors of Outcome

## Lead Researcher: Constantinos Sofocleous, MD, PhD [212-639-3379]

If you are the parent or legal guardian of the person who is being asked to participate in this research study, you may give consent on his or her behalf. The word "you" in this document refers to your child, if the participant is a minor, or to a person with a cognitive impairment for whom you are the Legally Authorized Representative (LAR).

## **Overview and Key Information**

## Why is this study being done?

We are asking you to take part in a clinical research study. We do research studies to try to answer questions about how to prevent, diagnose, and treat diseases like cancer.

The treated tumor is normally evaluated with CT. The CT shows signs of treated tumor(s) in the area treated by ablation. However, cancer cells may begin to grow in or near the treated area. The CT scan cannot tell us if the cells are new cancer cells or if they are healthy liver cells that just look different because of the ablation. The test we will study should be able to tell us the difference.

## Taking part in this study is your choice.

You can choose to take part or not to take part in this study, and you can change your mind at any time. Whatever choice you make, you will not lose access to your medical care or give up any legal rights or benefits.

This document presents important information to help you make your choice. Please take time to read it carefully. Talk with your doctor, family, or friends about the risks and benefits of taking part in this study. It's important that you have as much information as you need, and that all your questions are answered.

## What is the usual approach to my cancer?

You will be having percutaneous ablation for tumor(s) that spread into your liver. The purpose of this study is to see if we can do some tests on tissue from the area of the ablation. We want to know if a test can help predict whether the ablation worked.

## What are my other choices if I decide not to take part in this study?

- You may choose to have the usual approach described above
- You may choose to take part in a different research study, if one is available
- You may choose not to be treated for cancer
- You may choose not to be treated for cancer, but to receive comfort care to help relieve your symptoms

# What will happen if I decide to take part in this study?



You will be asked to allow us to follow your results and image studies for 3 years after your treatment.

As part of your standard of care treatment for your cancer, you will be asked to return to clinic for follow up approximately 4-8 weeks after your percutaneous ablation procedure and approximately every 2-4 months for 3 years after.

## What are the risks and benefits of taking part in this study?

There are both risks and benefits to taking part in this study. It is important to think carefully about these as you make your decision.

#### Risks

We want to make sure that you know about a few key risks right now. We will also give you more information in the *What risks can I expect from taking part in this study?* section of this consent form.

If you choose to take part in this study, there is a risk that the percutaneous ablation may not be as good as CT scan at showing signs of treated tumor(s).

There is also a risk that you could have side effects from the percutaneous ablation. These side effects may be worse, and they may be different than you would have with the usual approach for CT.

Some of the most common side effects that the study doctors know about are:

- Bleeding
- Skin Burns

There may be some risks that the study doctors do not yet know about.

#### **Benefits**

Taking part in this study may or may not make your health better. We do know that the information from this study will help doctors learn more about percutaneous ablation as a treatment for cancer. This information could help future cancer patients.\

## If I decide to take part in this study, can I stop later?

Yes, you can decide to stop participating in the study at any time.

The study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

If you decide to stop, let the study doctor know as soon as possible. It's important that you stop safely.

If you stop, you can decide whether to let the study doctor or a member of the study team continue to contact you to ask questions about your health. We will not be able to withdraw information about you that has been used or shared with others before you informed us of your decision to stop.

## Are there other reasons why I might stop being in the study?

Yes. The study doctor may take you off the study if:

- Your health changes, and the study is no longer in your best interest
- New information becomes available, and the study is no longer in your best interest



- You do not follow the study rules
- The study is stopped by the Institutional Review Board (IRB), Food and Drug Administration (FDA), or the study sponsor, MSKCC. The study sponsor is the organization that oversees the study.

It is important that you understand the information in this informed consent document before you make a decision about participating in this clinical trial. Please read, or have someone read to you, the rest of this document. If there is anything that you don't understand, ask the study doctor or nurse for more information.

## What is the purpose of this study?

About 160 people will take part in this study at Memorial Sloan Kettering Cancer Center (MSK).

## What extra tests and procedures will I have if I take part in this study?

### Before you begin the main part of the study:

The study doctor will review your medical records and the results of your exams, tests, and procedures to see if it is safe for you to take part in the study. This first part of the study is called screening. Most of the screening exams, tests, and procedures are part of the usual care that you would have if you were not in a study.

The tests and procedures that will be done only for research purposes, or that may be done more often because you are participating in this study, are listed below.

These things will be done whether you choose to be part of the study or not. It is part of the normal work-up for all patients that undergo percutaneous ablation of liver tumors:

Approximately within 30 days of the percutaneous ablation procedure you will have a:

- Office visit with the interventional radiologist who will do the percutaneous ablation
- Blood test (the blood tests will let us know if you can safely have the percutaneous ablation treatment)
- A CT of the chest, abdomen and pelvis. This CT imaging test is done before and after the injection of X-ray dye through an IV line. (If the contrast dye that is used in the CT scan is not indicated for you, you will have an MRI scan instead).
- Recommended whole Body PET/CT, as per your standard of care

#### **During the study:**

 Your tumor will be treated using percutaneous ablation according to the standard care for your cancer. The percutaneous ablation will be guided by the CT scanner or PET/CT scanner. Collection and testing of tissue if found on the percutaneous ablation device

#### Exams, Tests and/or Procedures

You will have procedures during the main study. The procedures that will be done only for research purposes, or that may be done more often because you are participating in this study, are listed below.

- Biopsy of the tumor(s) before ablation treatment
- Biopsy of the tumor(s) after the ablation treatment
- Testing of the tissue collected by the biopsy



# Memorial Sloan Kettering Cancer Center IRB Number: 09-122 A(22)

Approval date: 12-Apr-2022

During your image-guided percutaneous ablation, you will be put to sleep and monitored by an anesthesiologist. You will have a CT without contrast to focus on the liver tumor that will be treated. After the tumor is found with the CT, the Interventional Radiology doctor will place a needle and take tissue then perform the percutaneous ablation. Right after the percutaneous ablation, you will have a CT with contrast to make sure all of the tumor was destroyed. Before the CT, you will have a needle placed into the vein in your arm. This is called intravenous or IV. This is for injecting contrast into your arm. The contrast helps the doctor interpret the CT scan.

The IR doctor will use the CT images to place a needle inside the destroyed tumor. Tissue will be taken through the needle. The needle is usually placed through the same hole as the ablation needle. We will send the tissue to our lab for the testing.

Once the testing is done, you will go to the post-anesthesia to recover. You will stay there overnight so the nurses can watch you. This is standard for percutaneous ablation. You will stay there whether or not you take part in this study.

If as part of your standard of care treatment the doctor feels that you must be retreated with another percutaneous ablation, the ablation will be repeated as previously described. A new biopsy and testing of tissue will be done from the area of the repeated ablation. The goal of the biopsy is to detect if there are any cancer cells left behind in the area that was treated with percutaneous ablation. All biopsies, tissue collections and lab evaluations will be exactly the same after each ablation as described.

### **End-of-Treatment and follow-up visits:**

This follow-up will be performed whether you choose to be part of the study or not. It is part of the standard follow-up for all patients that have percutaneous ablation of liver tumors. After you are finished with the study, the study doctor will ask you to have:

- There will be a follow up phone conversation approximately 1-2 weeks after treatment to determine your recovery. If you have not fully recovered and are experiencing difficulties, you will be instructed to see a doctor. If you are unable to come to MSKCC to do blood work and have a physical examination, it will be necessary to see your local doctor and to have the blood work done locally. These results will have to be faxed to the IR doctor that treated you.
- Follow up visits after percutaneous ablation will include: CT of the chest, abdomen and pelvis with IV x-ray dye and PET/CT approximately 4-8 weeks after your percutaneous ablation procedure and then approximately every 2-4 months thereafter.
- Standard Care Blood tests. Blood tests after percutaneous ablation are performed to make sure that there is no injury to your liver after treatment. Blood tests are also done to keep an eye on tumor markers such as CEA in patients with colon cancer. If your CEA level was high before the procedure, you will be instructed to have a CEA level drawn either at MSKCC or at your local hospital approximately 1-2 weeks after percutaneous ablation, and again approximately 4-8 weeks after percutaneous ablation and then approximately every 2-4 months for three years.



### Will I receive the results of my research tests?

Neither you nor your doctor will receive the results of any tests done for research purposes during this study.

## What risks can I expect from taking part in this study?

If you choose to take part in this study, there is a risk that:

- You may lose time at work, school, or at home, and you may spend more time than usual in the hospital or doctor's office
- You may be asked sensitive or private questions that you do not usually discuss

The percutaneous ablation used in this study may affect how different parts of your body work, such as your liver, kidneys, heart, and blood. The study doctor will be testing your blood throughout the study, and he or she will let you know if changes occur that may affect your health.

There is also a risk that you could have side effects from the study drug(s)/study approach.

Important information about side effects:

- The study doctors do not know who will or will not have side effects.
- Some side effects may go away soon, some may last a long time, and some may never go away.
- Some side effects may make it difficult for you to have children.
- Some side effects may be mild. Others may be very serious and may even result in death.

Important information about how you and the study doctor can make side effects less of a problem for you:

- If you notice or feel anything different, tell the study doctor. He or she can check to see if you are having a side effect.
- The study doctor may be able to treat some side effects.
- The study doctor may adjust the study drugs to try to reduce your side effects.

The tables below show the most common and the most serious side effects that researchers know about. There may be other side effects that the doctors do not yet know about. If important new side effects are found during this study, the study doctor will discuss them with you.

#### Possible side effects of Percutaneous Ablation:

#### Common, some may be serious

In 100 people receiving Percutaneous Ablation, more than 20 and as many as 100 may have:

Immediate complications are bleeding. Most of the time a small amount of blood in the
area where the tumor was treated is seen. The bleeding usually stops and there are
no symptoms and no more treatment is required.

### Occasional, some may be serious

In 100 people receiving Percutaneous Ablation, between 4 and 20 may have:

• Collapsed Lung: If the tumor is located in an area close to the lung, there is a possibility that the needle used during the percutaneous ablation will prick the lung and cause some air to escape. This is called a collapsed lung. It happens in some



Occasional, some may be serious

In 100 people receiving Percutaneous Ablation, between 4 and 20 may have: patients when the needle goes through the lung. If this happens, the IR doctor doing the procedure will treat you right away. He/she will place a small tube around the lung. This will empty the air that is leaking from the hole in the lung.

#### Rare, and serious

In 100 people receiving Percutaneous Ablation, 3 or fewer may have:

- Severe bleeding. Although this is very rare, if this happens, it will be treated with blood transfusions or by embolization. Embolization is a procedure done by your IR doctor in order to find and close the vessel that was injured and caused the bleeding.
- Spreading of tumor along the path of the needle is a very serious side effect. It is an extremely rare complication (less than one in 100).
- Skin burns. This is a very rare complication. It occurs in less than one in 100. It
  happens at the area of the percutaneous ablation machine grounding pads or at the
  area where the needle enters the skin. Both are usually heal themselves or are
  treated with medical treatment. Specifically, if you are treated with IRE ablation, this
  may affect your normal heartbeat. The IR doctor will coordinate the electrical pulses
  used for this treatment method with information about your cardiac function during
  the procedure to minimize this risk.
- Bleeding that can be caused by the needle used in the biopsies to obtain tissue from your tumor. Most of the time bleeding after the biopsy stops and causes no symptoms. If a lot of bleeding happens after the needle biopsy, it will be treated with a blood transfusion or embolization.

Let the study doctor know about any questions you may have about possible side effects. You can ask the study doctor questions about side effects at any time.

## What are my responsibilities in this study?

If you choose to take part in this study, you will need to:

- Keep your study appointments
- Tell the study doctor about:
  - All medications and any supplements you are taking
  - Any side effects from these medications or supplements
  - Any doctor visits or hospital stays outside of this study
  - Whether you have been or are currently in another research study

## Is there a conflict of interest for this study?

This study is sponsored by Memorial Sloan Kettering Cancer Center

No conflicts of interest have been identified for either the institution or the investigator(s) in this study.



# What are the costs of taking part in this study?

You will not have to pay for the percutaneous ablation or for tests and procedures done only for research purpose.

It is possible that ablation may not continue to be supplied while you are in the study. This possibility is unlikely, but if it occurs, your study doctor will talk with you about your options.

You and/or your health plan/insurance company will have to pay for all the other costs of treating your cancer while you are in this study. These charges include the costs of insurance co-pays and deductibles, as well as tests, procedures, or drugs that you get during the study to monitor your safety, and to prevent or manage any side effects.

Talk to your insurance provider and make sure that you understand what your insurance pays for and what it does not pay for if you take part in this clinical trial. Also find out if you need approval from your health plan before you can take part in this study.

The study doctor or nurse can help you find the right person to talk to if you are not sure which costs will be billed to you or your insurance provider.

## Will I receive payment for taking part in this study?

You will not be paid for taking part in this study.

## What happens if I am injured or hurt because I took part in this study?

You will get medical treatment if you are injured as a result of taking part in this study.

If you think that you have been injured as a result of taking part in this research study, tell the study doctor or the person in charge of the study as soon as possible. The name and telephone number of the person in charge of this research are listed on the first page of this consent form.

We will offer you treatment for research injuries that happen as a result of your taking part in this study. You and/or your health plan will be charged for this treatment. Medical services will be offered at the usual charge. You will be responsible for any costs not covered by your health plan/insurance company. If you think that your injury was a result of medical error, you keep all your legal rights to receive payment for treating the injury, even though you are in a study.

## Who will see my medical information?

Your privacy is very important to us, and the researchers will make every effort to protect it. Trained staff at Memorial Hospital may review your records, if necessary.

Access to your protected health information will be limited to those listed in the Research Authorization form, which is a part of the informed consent process.

Your information may be given out, if required by law. For example, some states require doctors to make a report to the state health board if they find that a participant in a research study has a contagious disease like tuberculosis. However, the researchers will do their best to make sure that any information about you that may be released will not identify you.



### Memorial Sloan Kettering Cancer Center IRB Number: 09-122 A(22) Approval date: 12-Apr-2022

In the future, your information (data) may be de-identified, which means that your data will be assigned a unique code, and the list that links the code to your name will be stored separately from your data. Your de-identified information may be used for research that has not been described in this consent form, and they may be shared with another investigator for future research. You will not be asked if you agree to take part in future research studies.

If your information from this study is used in any reports or publications, your name and anything else that could identify you will not be used. It is possible that your de-identified information from this study will be shared with other researchers outside of MSK and may be stored in public databases. All requests for data sharing will be reviewed by the study sponsor, and if individual results are included in the data, they will not contain any identifiable information about you, such as your name, address, telephone number, or social security number. Your privacy is very important to us and we use many safety procedures to protect your privacy. However, we cannot guarantee that no one will ever be able to use your information to identify you.

Some of your health information and/or information about your specimens from this study will be kept in a central database for research. Your name and contact information will not be stored in the database.

The study doctors have certified a Certificate of Confidentiality from the National Institutes of Health for this study. This gives MSK an additional way to protect sensitive information that identifies you in your records if it is requested as part of a legal proceeding. However, MSK may still be required to share some of your medical information if required by law.

## Where can I get more information?

You may visit the NCI web site at <a href="http://cancer.gov/">http://cancer.gov/</a> for more information about research studies, or for general information about cancer. You may also call the NCI Cancer Information Service to get the same information at 1-800-4-CANCER (1-800-422-6237).

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

You can talk to the study doctor about any questions or concerns that you may have about this study, or to report side effects or injuries. You may also contact the lead researcher listed on the first page of this consent.

For questions about your rights while you are participating in this study, call the MSK Institutional Review Board (IRB) at 212-639-7592. If you have concerns, complaints, or input on research, or if you would like more information about the informed consent process, please contact the MSK Patient Representative Department at 212-639-7202.



# Research Authorization for the Use and Disclosure of Protected Health Information (PHI)

Examinations of Tissue from Ablated Malignant Liver Metastases as Predictors of Outcome

Federal law requires Memorial Sloan Kettering Cancer Center (MSK) to protect the privacy of information that identifies you and relates to your past, present, and future medical conditions (protected health information; PHI). We are committed to protecting the privacy of your information.

If you enroll in this research study, your protected health information will be used and shared with others, as explained below. MSK must obtain your permission before using or sharing your protected health information for research purposes. This form helps to make sure that you are informed of the ways in which your information will be used or shared in the future.

Carefully read the information below before you sign this form. By signing this form, you agree to the use and disclosure of your information for this research study.

# 1. What protected health information about me will be used or shared with others during this research?

- Your medical records
- Your research records, including new health information created from study-related tests, procedures, visits, and/or questionnaires
- HIV-related information, including any information indicating that you have had an HIV-related test; or that you have HIV infection, HIV-related illness, or AIDS; or any information that could indicate that you may have been exposed to HIV. (New York State requires us to obtain your consent to use or share this information.)

## 2. Who will use or share my protected health information?

MSK will use and share your protected health information. People and offices that deal with research oversight, quality assurance, and/or billing will be able to use and share your protected health information, including:

- The study's Principal Investigator and Co-Principal Investigator(s): Constantinos Sofocleous, MD, PhD; and Katia Manova PhD;
- Your research team at MSK, including the participating investigators, research staff, research nurses, fellows/residents, and clerical support staff
- Any healthcare personnel who provide services to you in connection with this study
- Members and staff of MSK's Institutional Review Board (IRB) and Privacy Board (PB)
- Staff of MSK's Clinical Research Administration, which oversees clinical studies, and Clinical Research Information Technology Group, which manages research databases
- Members of MSK's Data Safety Monitoring Board/Committee and the Quality Assurance Committee



# 3. With whom outside of MSK may my protected health information be shared?

Although all reasonable efforts will be made to maintain the confidentiality of your protected health information, it may be shared with and used by the following:

- MSK's research collaborators, business partners, subcontractors and agent(s), in the United States or in other countries, working to conduct the study, to monitor the study, or to analyze the study information for this study or for other research about the study procedure.
- Other research doctors and medical centers participating in this research.
- Federal and state agencies, and other domestic or foreign government bodies, if required by law and/or necessary for oversight purposes, including:
  - Office for Human Research Protections (OHRP) of the US Department of Health and Human Services (HHS)
  - US Food and Drug Administration (FDA) and other regulatory agencies responsible for oversight of research
  - National Cancer Institute (NCI)/National Institutes of Health (NIH)

Some of the organizations that may receive your protected health information may not have to satisfy the privacy rules and requirements; they may share your information with others without your permission.

# 4. Why will my protected health information be used by or shared by MSK or others?

The main reasons for the use or sharing of your information include the following:

- To conduct the study, to monitor your health status, to measure the effects of the drug(s)/device(s)/procedure(s) being studied, and to determine the research results
- To ensure that the research meets legal and institutional requirements
- To develop new tests, procedures, and commercial products
- To enhance research databases, so that scientists can design better research studies to develop new therapies for patients and to gain a better understanding of disease
- To assist with MSK medical treatment, billing, or healthcare operations. For example, medical information produced by this research study will become part of your hospital medical record.

# 5. For how long will my protected health information be used or shared with others?

There is no set date at which your protected health information that is being used or shared for this research study will be destroyed or no longer used. The information used and created during the study may be analyzed for many years, and it is not possible to know when this analysis will be completed.



## 6. Statement of privacy rights:

- It is your right to refuse to sign this authorization form. If you do not sign this form, you will not be able to participate in this research study. However, if you do not sign, it will not affect your ongoing medical treatment or healthcare coverage.
- You have the right to withdraw your permission for MSK to use or share your protected health information. Please note that we will not be able to withdraw all the information about you that already has been used or shared with others to carry out research-related activities such as oversight, or information that is needed to ensure the quality of the study. To withdraw your permission, write to the study doctor listed on the first page of this consent form at: Memorial Sloan Kettering Cancer Center, 1275 York Avenue, New York, NY 10065. If you withdraw permission for us to use or share your protected health information, you will not be able to continue to participate in this research study.
- You have the right to request access to your protected health information that is being used or shared during this research and that is related to the research or to payment for the research. However, you may access this information only after the study is completed. You may have access to your medical record at any time. To request this information, please contact the study doctor whose name and telephone number are listed on the first page of this consent form. You may also ask the study doctor to correct any study-related information about you that is wrong.

### **Notice concerning HIV-related information**

Individuals/organizations are prohibited from sharing any HIV-related information about you without your approval, unless they are permitted to do so under federal or state law. You have a right to request the list of people who may receive or use your HIV-related information without your authorization.

If you experience discrimination because of the release or disclosure of your HIV-related information, you may contact the New York State Division of Human Rights at 888-392-3644 or the New York City Commission on Human Rights at 212-306-7500. These agencies are responsible for protecting your right

# Participant Informed Consent/Research Authorization for Clinical Research

#### Statement of professional obtaining consent

I have fully explained this clinical research study to the participant or to his/her Legally Authorized Representative (LAR). In my judgment, and in that of the participant or his/her LAR, sufficient information



Memorial Sloan Kettering Cancer Center IRB Number: 09-122 A(22)

Approval date: 12-Apr-2022

including risks and benefits, was provided for the participant or his/her LAR to make an informed decision. The consent discussion will be documented in the participant's EMR.

| Consenting profess | sional must personally sign and | l date |
|---|---|---|
| Consenting professional's | | Date: |
| signature Consenting professional's name | | |
| (Print) | | |

#### Participant's (or Legally Authorized Representative's [LAR's)]) statement

I have read this form that describes the clinical research study. I have also talked it over to my satisfaction with the consenting professional. By signing below, I agree to the following: (1) to voluntarily participate in this clinical research study; (2) to authorize the use and dis

closure of my/the participant's protected health information (data about myself/the participant); and (3) to state that I have received a signed and dated copy of this consent form.

| nally sign and date |
|---------------------|
| Date: |

| Witness signature (if required) | |
|---|---|
| | Witness for non-English speaking participant: I declare that I am fluent in both English and in the |
| | participant's (or LAR's) language, and I confirm that the consent discussion was appropriately interpreted |
| | for the participant (or LAR). |
| | ☐ Other: I confirm that the consent discussion occurred, and that the participant agreed to participate in |
| | this study by signing this form, making his/her mark, or verbally agreeing. |
| Name of witness: | |
| Si | gnature of witness: Date: |
| (Tł | ne name of the witness must be documented in the EMR.) |
| In | terpreter (if required) |
| Na | me of interpreter (if present): |
| ID number (if phone interpreter): | |
| (Tł | (The interpreter's name or ID number must be documented in the EMR.) |

The participant/Legally Authorized Representative must be provided with a **signed copy** of this form.

